CLINICAL TRIAL: NCT03092947
Title: Use of Preoperative Renal Functional Reserve to Predict Risk of Acute Kidney Injury After Cardiac Surgery
Brief Title: Preoperative Prediction of Acute Kidney Injury After Cardiac Surgery
Acronym: RFR
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Faeq Husain, Senior Physician, University of Giessen
Other Study IDs: n63/14
Record Dates: First submitted 2017-03-21; First posted 2017-03-28 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of only residual material (blood, urine) for International Renal Research Institute
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Although acute kidney injury (AKI) frequently complicates cardiac surgery, methods to determine AKI risk are lacking. Renal functional reserve (RFR), the capacity of the intact nephron mass to increase glomerular filtration rate (GFR), represents maximal filtration capacity. We hypothesized that preoperative RFR would predict postoperative AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a frequent complication in patients undergoing cardiac surgery with an estimated prevalence of 36%. However, clinicians have limited tools to preoperatively identify patients at risk for AKI and/or progression to chronic kidney disease, particularly in patients with normal resting glomerular filtration rate (rGFR). Renal functional reserve (RFR) describes the capacity of the intact nephron mass to increase GFR from baseline in response to stimuli (e.g., protein load). We hypothesized that the presence or absence of RFR could separate patients at risk for developing AKI from patients with better-preserved renal function and a more favorable short- and long-term prognosis despite identical rGFR. The aim of this study is to examine whether preoperative assessment of RFR is able to predict risk for AKI after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects older than 18 years
2. Subjects undergoing elective cardiac surgery
3. Subjects who signed informed consent forms

Exclusion Criteria:

1. Pregnancy
2. Chronic kidney disease ≥ stage III
3. Solitary kidney
4. Diabetes mellitus type 1
5. Recent cardiac arrest
6. Liver failure or cirrhosis
7. Total parenteral nutrition
8. Hemoglobin <11 g/dl
9. Sepsis
10. History of malabsorption, chronic inflammatory bowel disease, short bowel, or pancreatic insufficiency
11. Transplant donor or recipient
12. Active autoimmune disease with renal involvement
13. Rhabdomyolysis
14. Prostate hypertrophy with International Prostate Symptom Score ≥20
15. Neoplasm

Withdrawal criteria:

All patients included in the study were to be followed up until the scheduled end of the study. Data collection could be terminated prior to the scheduled time only under the following conditions:

* General criteria

  1. A patient or his/her legal representative may refuse further participation in the study at any time (withdrawal of consent),
  2. The investigator may withdraw a patient from the participation in the study at any time for the following reasons:

     * a severe protocol violation,
     * the development of incidents/near-incidents/other severe clinical complications related to the study protocol
* Criteria related to the study

  1. Subjects who could not stop taking angiotensin-converting enzyme inhibitors and/or angiotensin II receptor blockers a minimum of 48 hours before the protein load.
  2. Subjects who received non-steroidal anti-inflammatory drugs within the 48 hours before the protein load.
  3. Subjects who received intravenous radiocontrast agents within the 72 hours before the protein load.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
The predictive value of RFR for AKI in patients undergoing elective cardiac surgery | 1 day before cardiac surgery

SECONDARY OUTCOMES:
Whether the occurrence of AKI (as defined by Kidney Disease Improving Global Outcomes criteria) impacts RFR three months after surgery in patients without ongoing reduced function defined by resting GFR | 3 months after cardiac surgery
Whether urinary [TIMP-2][IGFBP7] predicts loss of RFR | 3 months after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, MD, Study Director — International Renal Research Institute of Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haase M, Kellum JA, Ronco C. Subclinical AKI--an emerging syndrome with important consequences. Nat Rev Nephrol. 2012 Dec;8(12):735-9. doi: 10.1038/nrneph.2012.197. Epub 2012 Sep 25. PMID 23007617
- [Result] Sharma A, Zaragoza JJ, Villa G, Ribeiro LC, Lu R, Sartori M, Faggiana E, de Cal M, Virzi GM, Corradi V, Brocca A, Husain-Syed F, Brendolan A, Ronco C. Optimizing a kidney stress test to evaluate renal functional reserve. Clin Nephrol. 2016 Jul;86(7):18-26. doi: 10.5414/CN108497. PMID 27285313
- [Result] Ronco C, Chawla LS. Glomerular and Tubular Kidney Stress Test: New Tools for a Deeper Evaluation of Kidney Function. Nephron. 2016;134(3):191-194. doi: 10.1159/000449235. Epub 2016 Aug 30. PMID 27577054
- [Derived] Husain-Syed F, Emlet DR, Wilhelm J, Danesi TH, Ferrari F, Bezerra P, Lopez-Giacoman S, Villa G, Tello K, Birk HW, Seeger W, Giavarina D, Salvador L, Fuhrman DY, Kellum JA, Ronco C; IRRIV-AKI Study Group. Effects of preoperative high-oral protein loading on short- and long-term renal outcomes following cardiac surgery: a cohort study. J Transl Med. 2022 May 10;20(1):204. doi: 10.1186/s12967-022-03410-x. PMID 35538495
- [Derived] Husain-Syed F, Ferrari F, Sharma A, Hinna Danesi T, Bezerra P, Lopez-Giacoman S, Samoni S, de Cal M, Corradi V, Virzi GM, De Rosa S, Mucino Bermejo MJ, Estremadoyro C, Villa G, Zaragoza JJ, Caprara C, Brocca A, Birk HW, Walmrath HD, Seeger W, Nalesso F, Zanella M, Brendolan A, Giavarina D, Salvador L, Bellomo R, Rosner MH, Kellum JA, Ronco C. Persistent decrease of renal functional reserve in patients after cardiac surgery-associated acute kidney injury despite clinical recovery. Nephrol Dial Transplant. 2019 Feb 1;34(2):308-317. doi: 10.1093/ndt/gfy227. PMID 30053231
- [Derived] Husain-Syed F, Ferrari F, Sharma A, Danesi TH, Bezerra P, Lopez-Giacoman S, Samoni S, de Cal M, Corradi V, Virzi GM, De Rosa S, Mucino Bermejo MJ, Estremadoyro C, Villa G, Zaragoza JJ, Caprara C, Brocca A, Birk HW, Walmrath HD, Seeger W, Nalesso F, Zanella M, Brendolan A, Giavarina D, Salvador L, Bellomo R, Rosner MH, Kellum JA, Ronco C. Preoperative Renal Functional Reserve Predicts Risk of Acute Kidney Injury After Cardiac Operation. Ann Thorac Surg. 2018 Apr;105(4):1094-1101. doi: 10.1016/j.athoracsur.2017.12.034. Epub 2018 Jan 31. PMID 29382510